CLINICAL TRIAL: NCT04263428
Title: The Effects of Sleep Variability on Sleep Quality, Daytime Functioning and Cardiometabolic Regulation in Youth
Brief Title: The Effects of Sleep Variability in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Director of the Sleep Research Clinic and Laboratory, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EA1708030
Record Dates: First submitted 2019-06-15; First posted 2020-02-10 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Sleep Variability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irregular sleep (Experimental): Participants sleep in lab while being monitored with polysomnography for 8 consecutive nights, including an adaptation night and a baseline night of 7.5 h time in bed (0:00-7:30). Afterwards, they are instructed to sleep in bed on a schedule alternated between 6 h, i.e. 1:30-7:30, and 9 h, i.e. 22:30-7:30).
  Interventions: Behavioral: Irregular sleep
- Regular sleep (No Intervention): Participants sleep in lab while being monitored with polysomnography for 8 consecutive nights of 7.5 h time in bed (0:00-7:30).

INTERVENTIONS:
Behavioral: Irregular sleep — Experimental-induced sleep variability
  Arms: Irregular sleep

SUMMARY:
Daily sleep variability is prevalent in the young populations, yet its effects remain less clear. The experimental study aims to examine the impacts of intraindividual daily sleep variability on sleep characteristics, cardiometabolic regulations and daytime functioning in college students.

ELIGIBILITY:
Inclusion Criteria:

* Habitual sleep duration > 7 h/day.

Exclusion Criteria:

* Extreme morning- nor extreme evening-chronotype
* With sleep problems
* With mood and anxiety problems
* With excessive daytime sleepiness
* Have history of any chronic medical condition and on regular medication.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Subjective sleepiness | 7 days (every morning and evening)
  As measured by the Stanford Sleepiness Scalen (SSS)
Mood | 7 days (every morning and evening)
  mood state as measured by the Positive and Negative Affect Scale (PANAS).
Cognitive functioning - Sustained attention | 7 days (every morning and evening)
  Sustained attention as measured by psychomotor vigilance task (PVT)
Cognitive functioning - processing speed | 7 days
  Processing speed as measured by Digit Symbol Substitution Test (DSST)
Cognitive functioning - inhibition | 7 days
  Inhibition as measured by stop-signal reaction time (SSRT)
Cognitive functioning - working memory | 7 days
  working memory as measured by 2-back task

SECONDARY OUTCOMES:
Sleep quality | 7 days
  Actual sleep time, sleep onset latency, wake after sleep onset and night time arousals as measured by actigraphy and PSG. Sleep satisfactory and dreams as measured by sleep diary.
Sleep architecture | 7 days
  Sleep stagings (e.g., SWS%, REM duration) and sleep EEG spectrums as analysed from PSG recordings.
Heart rate variability | 7 days
  Resting heart rate and heart rate variability are measured in the morning, evening and during the night.
Cortisol awakening response | baseline, post-intervention
  Cortisol awakening response is assessed before and after the manipulation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shirley X. Li, Principal Investigator — The University of Hong Kong
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong